CLINICAL TRIAL: NCT00610246
Title: A Phase I Dose Escalation Study of Concurrent Low Dose Radiation With Sorafenib in Three Anatomically-based Independent Cohorts (Thorax, Abdomen, Pelvis)
Brief Title: A Study of Radiation With Sorafenib in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAP; DDPDRO-003 (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cancer
Keywords: Thorax; Abdomen; Pelvis; Lesion; Cancer; Radiation; Chemotherapy; Phase 1; Advanced Cancer; Sorafenib; Nexavar; BAY43-9006
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and Radiation (Experimental): Eligible patients (not candidates for curative treatment) will have measurable lesions in the anatomic thorax, abdomen or pelvis (any histology) amenable to palliative radiation treatment (30 Gy in 10 fractions). Patients receive sorafenib orally for one week prior to radiation, then concomitantly for two weeks with radiation and then for one week following completion of radiation. Each anatomic cohort will dose escalate independently. If full oral dose (400 mg po bid) is reached in a given cohort (dose level three) then an additional dose level will open where sorafenib treatment (400 mg bid) is extended following radiation for a total of eight weeks.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib orally for one week prior to radiation, then concomitantly for two weeks with radiation and then for one week following completion of radiation. Each anatomic cohort will dose escalate independently. Dose level 1 is 200mg of sorafenib. If full oral dose (400mg orally, twice a day) is reached in a given cohort then an additional dose level will open where sorafenib treatment is extended following radiation for a total of eight weeks.

SUMMARY:
The purpose of this study is to test the combination of radiation treatment and an anti-angiogenic drug called sorafenib (or BAY 43-9006 or Nexavar) to determine the effects of this combination on cancers but also on side effects of radiation treatment. This study will also determine the highest safe dose of sorafenib that can be given with radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer not eligible for curative treatment.
* A measurable lesion in the thorax, abdomen or pelvis.
* Normal organ and bone marrow function.
* Able to receive protocol prescribed radiation. Please refer to the protocol for detailed inclusion criteria.

Exclusion Criteria:

* Overlap of treatment field with a previous radiation field.
* Inability to meet mandated normal tissue radiation dose constraints.
* Brain metastases (unless previously treated and controlled)
* Previous treatment with Sorafenib.
* Poorly controlled Hypertension.
* Unable to swallow sorafenib tablets.
* Intercurrent cardiac dysfunction.
* Uncontrolled intercurrent illness. Please refer to the protocol for detailed exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Outcome is measured prior to each dose escalation.
  To measure safety and maximum tolerated dose, all adverse events will be assessed in line with dose limiting toxicities.

SECONDARY OUTCOMES:
Sorafenib with radiation treatment efficacy | 12 weeks from initiation of study treatment.
  To assess the efficacy of adding sorafenib to radiation treatment, radiological imaging will be used to assess response rate inline with the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Brade, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada